CLINICAL TRIAL: NCT00404053
Title: One Year Effects of Different Clopidogrel Maintaining Dosage on Patients With Acute Coronary Syndrome Undergoing Coronary Drug Eluting Stent Implantation
Brief Title: Clopidogrel Maintaining Dosage in Acute Coronary Syndrome After Drug Eluting Stent Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH-2004-A003
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel

SUMMARY:
In view of its safety profile and the results of clinical trials, clopidogrel has become the standard treatment for patients with acute coronary syndrome (ACS) and drug eluting stent(DES) implantation. Two large studies in patients with ACS shown that pretreatment with clopidogrel had beneficial effects. The pretreatment regimens were given a mean of 6 days before intervention in the observational PCI-CURE trial and 3 to 24 h in the randomized CREDO trial respectively. Accordingly, current clinical practice carries out pretreatment with a 300mg loading dose of clopidogrel at least 6 h before DES implantation procedure in patients with ACS. Compared with the 300mg clopidogrel loading dose, 600mg loading dose exhibited a superior antiplatelet effect and improved short-term clinical outcomes in patients undergoing DES implantation for ACS according to recent a few publications. But despite clopidogrel 600mg loading dose and the routine use of 75mg per day as a maintaining dose, recurrent ischemic events occurred in some patients. Therefore, the goal of this study will evaluate the efficacy of a 600mg loading dose of clopidogrel plus 150mg per day as a maintaining dose in patients with ACS undergoing DES implantation.

ACS patients undergoing DES implantation who receive planned 600mg loading dose clopidogrel pretreatment are eligible for the study. All enrolled patients will be randomized to receive daily clopidogrel 75 mg or 150mg as maintaining doses starting as soon as post-PCI, in addition to daily aspirin 100 mg, and lasted for the first month after DES implantation. One month later, all patients receive daily clopidogrel 75mg until 9~12month after DES implantation. The primary endpoints include death of all causes, myocardial infarction, revascularization of the target lesson, sub-acute and late stent thrombosis one year after PCI, The secondary endpoints are major and minor bleeding events. The study will be powered to test the hypothesis that higher maintaining dose(150mg) of clopidogrel will reduce major adverse cardiac events compared to currently used common dose(75 mg) at one year following PCI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ACS and planned pretreatment with 600mg loading dose of commercially available clopidogrel (Plavix).
* between ages of 18 Years and above
* Presence of one or several stenosis in native coronary arteries requiring PCI and suitable for DES implantation.
* Willing and able to sign informed consent.

Exclusion Criteria:

* A history of bleeding diathesis.
* New York Heart Association functional class IV.
* Prior PCI or coronary bypass grafting < 3 months.
* contraindications to clopidogrel and aspirin (White blood cells counts < 4×109/L or platelet counts <100 g.l-1 ;creatinine clearance <25 ml • min-1 ;active liver disease).
* use of glycoprotein IIb/IIIa inhibitors before PCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Dr, Principal Investigator — Shenyang Northern Hospital